CLINICAL TRIAL: NCT02597088
Title: Development of Methods for Enhance Human Milk Presentation During Storage and Warming
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sharron Bransburg-Zabary Consulting services (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Sharron Bransburg-Zabary, Sharron Bransburg-Zabary, PhD IBCLC, Sharron Bransburg-Zabary Consulting services
Other Study IDs: 0156-15-SZMC
Record Dates: First submitted 2015-10-26; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-09

CONDITIONS: Human Milk, Breast Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Laboratory studies of the effect of human milk handling using a rage surface area bottle (study device) — Using laboratory studies of the effect of storage and heating on expressed human milk, the investigators will compare milk handled in regular bottle and bottle warmer and milk handled using the study device (large surface area bottle)

SUMMARY:
Human milk (HM) is more than a food complex; in addition to micronutrients and human-coded bioactive complexes it also includes many antioxidants, antibacterial, prebiotics, probiotics, immune-boosting constituents, and many other bioactive components. Some of these components may deteriorate during storage, and expressed EHM starts deteriorating as soon as it leaves the breast. Nevertheless, whenever nursing at the breast or feeding of fresh EHM is not possible, feeding of stored EHM is considered the next best thing to feeding at the breast. Efficient heat transfer abilities affect both heating and cooling processes.

In this study the investigators wish to test a new device that permits rapid heating and cooling processes. The investigators plan to measure some thermolabile constituents of HM in order to determine whether they might be protected by a more gentle warming process. The investigators plan to collect milk from mother, to mix it and to test the effect of storage and heating.

This experiment is design to test the feasibility and the efficiency of the device.

DETAILED DESCRIPTION:
Exclusive breastfeeding is the normative model against which all alternative feeding methods must be measured with regard to infant growth, health, development, and all other short and long-term outcomes.

Recommendations for what is "safe" storage of Expressed HM have been developed, mainly for use by HM banks, but what constitutes optimal storage is less evident. Optimal handling of Expressed HM (EHM) should include proper storage as well as proper heating and thawing prior to use, in order to reduce damage to its nutritional and bioactive components.

Efficient heat transfer abilities affect both heating and cooling processes. In a previous work , the investigators showed that overheating of EHM is highly probable when using commercially available electrical water-based bottle warmers, even if the manufacturer's recommendations are followed . Besides warming process, EHM stability can also be affected by container composition and shape, storage temperature and whether or not sterilization was effected prior to storage. Following our previous study, the investigators hypothesized that a non-standard storage and warming process may increase EHM preservation. The investigators therefore designed a novel device with larger surface area and narrower milk width in order to minimize temperature gradients within the milk volume.

The investigators plan to store and heat HM in regular baby bottle and in our device and test thermolabile properties of HM, such as certain proteins and microbiological cultures, to asses if the new device can indeed protect the milk.

In order to obtain EHM from mothers, the investigators will collected freshly pumped milk The pumped milk will be pooled into a single container. A milk samples will be taken to define the reference values then it will equally divide into three study containers and into six control containers (C-container, regular baby bottles). After filling, all containers will be placed in a dark refrigerator at the temperature of 4ºC.

The experiment will last for 5 days. On the first day, one S-container and two C-containers will be taken out of the refrigerator and tested: the milk in each container will be warmed to feeding temperature in the container; it was then stirred gently and a sample of the warmed milk was obtained and stored at -20ºC until analyzed. This procedure was repeated on days 3 and 5 of the experiment.

The warming procedure used on the C-containers was as follows: the C-container will be warmed in standard electric water-based bottle warmer. Usually the warmer has three heating options; fast, medium, and slow. Investigators plan to test the fastest option on three of the six bottles and the slowest option on the remaining three bottles. The heating process will be terminated once the temperature of the heated milk reached 37ºC.

The warming procedure used on the S-containers was as follows: the S-container was placed in a bowl containing water at approximately 40ºC and gently moved in circles until the EHM reached 37 ºC.

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding mother that can donate milk for the study

Exclusion Criteria:

* mothers that have milk supply issues

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Breastfeeding mothers. Up to 6 months PP. The milk will be mixed. The tested milk cannot be connected to specific donor.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Measurements of higher concentration of thermolabile proteins or/and higher activity level of thermolabile enzymes, in expressed human milk that was handled using the study device as compared to regular baby bottles | 3 months

SECONDARY OUTCOMES:
Less commensal bacterial growth measured using microbiological counts in the expressed milk that was handled using the study device as compared to regular baby bottles | 3 months
Faster warming time as in the study device compared with regular bottles. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharron Bransburg-Zabary, PhD, Principal Investigator — Consulting services